CLINICAL TRIAL: NCT00431132
Title: A 12 Month, Open-label, Multi-center Trial to Investigate the Endometrial Safety of Vagifem Low Dose (10ug 17beta-estradiol Vaginal Tablet) in Postmenopausal Women With Atrophic Vaginitis Symptoms
Brief Title: Endometrial Safety of a Low Dose of Vagifem® in Postmenopausal Women With Atrophic Vaginitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAG-1748; 2006-001629-24 (EudraCT Number)
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Menopause; Postmenopausal Vaginal Atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vagifem® 10 mcg (Experimental): One 10 mcg (microgram) vaginal tablet of intravaginal estradiol (Vagifem®) once daily for two weeks followed by one 10 mcg vaginal tablet twice weekly for 50 weeks
  Interventions: Drug: estradiol, 10 mcg

INTERVENTIONS:
Drug: estradiol, 10 mcg — Tablets, administered intravaginally twice weekly

SUMMARY:
This trial is conducted in Europe. The purpose of this study is to evaluate endometrial safety of intravaginal estradiol (Vagifem®) in healthy postmenopausal women having atropic vaginitis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women whose last menstruation was at least two years prior to the time of screening
* At least 1 urogenital symptom (vaginal dryness, vaginal and/or vulvar irritation/itching, vaginal soreness, dysuria, dyspareunia and vaginal bleeding associated with sexual activity
* Generally healthy

Exclusion Criteria:

* Exposure to exogenous sex steroid hormones (estrogen and/or progestin hormone replacement therapy) within past 3 months

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (34):
- Czechia (3):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Prague
- Denmark (6):
  - Novo Nordisk Investigational Site, Århus N
  - Novo Nordisk Investigational Site, Glostrup Municipality
  - Novo Nordisk Investigational Site, Herlev
  - Novo Nordisk Investigational Site, Hillerød
  - Novo Nordisk Investigational Site, Roskilde
  - Novo Nordisk Investigational Site, Virum
- Finland (5):
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- France (4):
  - Novo Nordisk Investigational Site, Évry
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Paris
- Hungary (3):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Pécs
  - Novo Nordisk Investigational Site, Szeged
- Norway (8):
  - Novo Nordisk Investigational Site, Drammen
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Larvik
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Sandvika
  - Novo Nordisk Investigational Site, Ski
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- Sweden (5):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Norrköping
  - Novo Nordisk Investigational Site, Uppsala

REFERENCES:
- [Result] Simon J, Nachtigall L, Ulrich LG, Eugster-Hausmann M, Gut R. Endometrial safety of ultra-low-dose estradiol vaginal tablets. Obstet Gynecol. 2010 Oct;116(4):876-883. doi: 10.1097/AOG.0b013e3181f386bb. PMID 20859151
- [Result] Simon J, Nachtigall L, Gut R, Lang E, Archer DF, Utian W. Effective treatment of vaginal atrophy with an ultra-low-dose estradiol vaginal tablet. Obstet Gynecol. 2008 Nov;112(5):1053-60. doi: 10.1097/AOG.0b013e31818aa7c3. PMID 18978105
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 sites in Czech Republic, Denmark, Finland, France, Hungary, Norway, and Sweden
Period: Overall Study
Arm/Group | Vagifem® 10 mcg
Started | 336
Completed | 292
Not Completed | 44

BASELINE CHARACTERISTICS:
Arm/Group | Vagifem® 10 mcg
Number analyzed (Participants) | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 336
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 296
  More than one race | 0
  Unknown or Not Reported | 39
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Endometrial Hyperplasia Based on Histological Assessment of Endometrial Biopsies
Description: The endometrial hyperplasia rate was calculated based on the number of patients with endometrial hyperplasia/endometrial carcinoma divided by the total number of subjects with interpretable biopsies at Week 52.
Time Frame: Week 52
Population: Safety analyses using LOCF (last observation carried forward) were performed on the safety population, which was comprised of 336 (100%) subjects who received 52 weeks of treatment with Vagifem® 10 mcg of trial drug.
Measure: Number; unit: percentage of participants
Arm/Group | Vagifem® 10 mcg
Number analyzed (Participants) | 336
percentage of participants
  Simple hyperplasia without atypia | 0
  Simple hyperplasia with atypia | 0
  Complex hyperplasia without atypia | 0
  Complex hyperplasia with atypia | 0
  Carcinoma | 0

2. Secondary Outcome: Transvaginal Ultrasound: Endometrial Thickness
Description: Transvaginal ultrasounds were performed at Baseline (Week 0) and Week 52, or at the time of withdrawal in the case of a subject's premature discontinuation. Endometrial thickness, measured (double layer) in mm, were lesser than 4 mm for entry into the trial.
Time Frame: Week 0, week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Vagifem® 10 mcg
Number analyzed (Participants) | 334
mm
  Baseline | 2.04 (0.9)
  Week 52 | 1.94 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a time frame of 12 months.
Description: Adverse events were collected from the first trial related activity after the subject has signed the informed consent to the end-of-trial. The safety population includes subjects who received 52 weeks of treatment with Vagifem 10 mcg of trial drug.
Arm/Group | Vagifem® 10 mcg
Serious Adverse Events (participants affected / at risk) | 14/336
Other Adverse Events (participants affected / at risk) | 17/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vagifem® 10 mcg (N=336)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vagifem® 10 mcg (N=336)
Nasopharyngitis (Infections and infestations) | 17 (18)

LIMITATIONS AND CAVEATS:
This was a single-arm, 12-month, open label, multicentre trial; therefore there were no comparator results available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication, or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.